CLINICAL TRIAL: NCT00473811
Title: Applicability of a Low Glycemic Index Diet in Diabetes
Brief Title: Diabetic Educational Eating Plan
Acronym: DEEP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Yunsheng Ma, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5P30DK032520-24 (NIH)
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Low-GI Dietary Education; ADA Dietary Education
Keywords: Glycemic index; carbohydrates; diabetes mellitus, type 2; randomized clinical trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADA diet (Active Comparator): Patients will be encouarged to consume foods consisted with ADA dietary recommendation
  Interventions: Behavioral: ADA diet
- Low-GI (Experimental): a low GI dietary education
  Interventions: Behavioral: Low GI

INTERVENTIONS:
Behavioral: Low GI — low-GI education
  Arms: Low-GI
Behavioral: ADA diet — ADA dietary education
  Arms: ADA diet

SUMMARY:
By improving glycemic control, many of the devastating complications of diabetes are to a large extent preventable. The use of a low GI (glycemic index) diet to improve glycemic control is relatively new and untested. However, a low GI diet may be a cost-effective approach to preventing diabetes-related complications. The aim of this proposed 2-year study is to gather pilot data on the feasibility of implementing a nutritionist-delivered low GI intervention, to reduce dietary GI in patients with type 2 diabetes, and to compare it with a nutritionist-delivered standard American Diabetes Association (ADA) diet intervention. Our outcomes are recruitment and retention rates, as well as physiological measures (HbA1c, blood lipids, blood pressure, and body mass index), dietary GI scores and acceptability of the intervention.

Primary hypotheses:

1. Recruitment and retention rates for the low GI intervention will be satisfactory.

Secondary hypotheses:

1. Participants in the low GI intervention group will show more favorable changes in physiological measures than participants in the ADA diet group.
2. Participants in the low GI group will be successful in lowering the GI of their diet.
3. Participants will find the intervention acceptable.

DETAILED DESCRIPTION:
The glycemic index (GI) is a ranking of carbohydrate containing foods according to the rate at which they raise blood glucose levels after eating. A recent meta-analysis of randomized clinical trials (RCT) suggests that choosing low GI foods has a small but clinically useful effect on medium-term glycemic control in patients with type 2 diabetes. However, in most of the reviewed RCTs, patients were fed experimental diets and therefore there is still controversy over the applicability of GI in the clinical setting for management of diabetes. In addition, there is no evidence that long-term consumption of a low GI diet will contribute to improved glycemic control in people with diabetes.

Our ultimate goal for a future larger RCT is to evaluate the long-term effects of using low GI diet in type 2 diabetics. The primary outcome variable of the future large trial will be glycosylated hemoglobin levels (HbA1c), a measure reflecting average glycemic level during the preceding 2-3 months. The proposed feasibility study will recruit 40 patients with type 2 diabetes and will randomly assign them to one of two groups: a low GI nutrition education group (low GI group) and a standard ADA dietary education group as the control group (ADA group) (20 patients in each group).

For both groups, the intervention phase will last 6 months and consist of an initial group session, an individual session, and then four group counseling sessions. The follow-up phase will be six months and consist of two group booster sessions, one at 8-months and another at 10-months. The low GI nutritional education will be primarily targeted at a low GI diet. The focus is not on decreasing total carbohydrate intake, but rather encouraging patients to substitute low GI foods for high GI foods. The dietary intervention will be based on a patient-centered counseling model which has been demonstrated to facilitate health behavior change. Data collection points coincide with two phases of the intervention. Assessments, including demographics, anthropometric measurements, diet and physical activity recalls, and clinical data, will be conducted at baseline, and at 6 and 12 months after randomization, with blood samples collected at each interval. We will track response to recruitment, adherence, and retention. Quantitative and qualitative methods will be used to assess acceptability of the intervention.

The aim of this proposed 2-year study is to gather pilot data on the feasibility of implementing a nutritionist-delivered low GI intervention to reduce dietary GI in patients with type 2 diabetes. Our outcomes are recruitment and retention rates, as well as physiological measures (HbA1c, blood pressure, and body mass index), dietary GI scores and acceptability of the intervention.

By improving glycemic control, many of the devastating complications of diabetes are to a large extent preventable. The use of a low GI diet to improve glycemic control is relatively new and untested. However, a low GI diet may be a cost-effective approach to preventing diabetes-related complications. Testing the feasibility of such a program and its potential impact would be an important step towards an RO1 application to the NIH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type II diabetes in the medical chart
* HbA1c level >= 7 (an indication of poor control of diabetes)
* Currently being treated with diet, oral hypoglycemic agents and/or insulin
* At least 21 years old
* Telephone in home or easy access to one
* Able to understand study protocol
* Understands and can provide informed consent
* Physician's approval to participate in study
* Has a blood glucose machine or a prescription for one from their physician
* Able to speak and read English
* Willing to be randomized to either of the two study groups
* Able to participate in the study for a one year length of time.

Exclusion Criteria:

* Pregnant or planning to become pregnant during the study
* Unable or unwilling to provide informed consent
* Plans to move out of the area within the 12-month study period
* Required intermittent glucocorticoid therapy within the past 3 months
* Documented acute coronary event (MI or unstable angina) within the past 6 months
* Diagnosis of a medical condition that precludes adherence to study dietary recommendations (e.g. Crohn's disease, ulcerative colitis, end-stage renal disease)
* Diagnosis of a psychiatric illness (i.e. dementia, psychiatric hospitalization or suicidality within the past 5 years). We will not exclude individuals with a diagnosis of depression or patients taking anti-depressants.
* Following a low-carbohydrate high fat dietary regimen such as the Atkins diet, or currently following the South Beach Diet
* Legally blind or has significant visual impairments

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Our outcomes are recruitment and retention rates, as well as physiological measures (HbA1c, blood pressure, and body mass index), dietary GI scores and acceptability of the intervention | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yunsheng Ma, MD, Ph.D., Principal Investigator — Division of Preventive & Behavioral Medicine, Department of Medicine, University of Massachusetts Medical School
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Ma Y, Olendzki BC, Hafner AR, Chiriboga DE, Culver AL, Andersen VA, Merriam PA, Pagoto SL. Low-carbohydrate and high-fat intake among adult patients with poorly controlled type 2 diabetes mellitus. Nutrition. 2006 Nov-Dec;22(11-12):1129-36. doi: 10.1016/j.nut.2006.08.006. Epub 2006 Oct 4. PMID 17027229
- [Result] Ma Y, Olendzki BC, Merriam PA, Chiriboga DE, Culver AL, Li W, Hebert JR, Ockene IS, Griffith JA, Pagoto SL. A randomized clinical trial comparing low-glycemic index versus ADA dietary education among individuals with type 2 diabetes. Nutrition. 2008 Jan;24(1):45-56. doi: 10.1016/j.nut.2007.10.008. PMID 18070658